CLINICAL TRIAL: NCT03950869
Title: The Role of Expectations in the Development of Intrusive Memories: An Experimental Approach Using the Trauma Film Paradigm
Brief Title: The Role of Expectations in the Development of Intrusive Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2019-07
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three arms in parallel for the duration of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Negative Expectations (Experimental): Expectations on the severity and frequency of intrusions are increased while expectations on the controllability of intrusions are decreased.
  Interventions: Behavioral: Negative Expectation Manipulation
- Positive Expectations (Experimental): Expectations on the severity and frequency of intrusions are decreased while expectations on the controllability of intrusions are increased.
  Interventions: Behavioral: Positive Expectation Manipulation
- No Expectation Manipulation (No Intervention): Expectations on the severity and frequency of intrusions and on the controllability are neither increased nor decreased.

INTERVENTIONS:
Behavioral: Positive Expectation Manipulation — Participants are watching a video tape of a trauma expert who provides selective information on the development of intrusive memories. This video tape aims to increase positive expectations.
  Arms: Positive Expectations
Behavioral: Negative Expectation Manipulation — Participants are watching a video tape of a trauma expert who provides selective information on the development of intrusive memories. This video tape aims to increase negative expectations.
  Arms: Negative Expectations

SUMMARY:
In the experimental study, the well-established trauma film paradigm will be used to investigate the impact of expectations on the development of intrusive memories as a hallmark symptom of PTSD.

DETAILED DESCRIPTION:
The study aims to examine the influence of different expectations on the development of intrusive memories by using a well-established experimental paradigm - the trauma film paradigm. In healthy volunteers, intrusion-like symptoms are to be induced with an analogue stressor, i.e., aversive film clip footage (trauma film). After viewing this so-called trauma film, the expectations of intrusions during the following week are manipulated by assigning participants randomly to three different groups. In the first group, negative expectations are induced (experimental group 1), the second group is exposed to positive expectations (experimental group 2) and a third group does not face any kind of manipulation of their expectations (control group). Participants are asked to report occurring intrusions in a diary during the following week and are invited to a subsequent cued laboratory inquiry at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* fluent in German language

Exclusion Criteria:

* history of traumatic experiences (LEC-5)
* presence of a mental disorder (SCID-I according to DSM-IV)
* cut-off in depression screening (PHQ-9)
* current suicidal thoughts/behavior or non-suicidal self-injury behavior (C-SSRS)
* medical history of heart disease or epilepsy
* history of fainting
* work experience in the medical field (e.g., nurses, paramedics, etc.)
* visual impairment
* students of psychology and medicine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of intrusive memories: Daily intrusion diary | Record of any intrusive memories of the trauma film content for Days 1 to 7 after the experimental manipulation.
  Participants are asked to complete a pen-and-paper diary 7 days in a row, reporting on intrusive memories in reference to the trauma film. They are asked to state the number of intrusions per day; each day of the diary is labeled and split into three sections (morning, afternoon, evening), and they are asked to mark in a box in the appropriate section when they experienced an intrusion. For each intrusion, they indicate the quality of the intrusion (image, thought or both), the intensity of and distress caused by the intrusion both on a scale ranging from 0 ("not at all") to 10 ("extremely"), the content of the intrusion, and the situation in which the intrusion occurred. Intrusive memory frequency across 7 days are calculated, whilst higher sum scores represent more intrusions. Severity of intrusions are calculated by combining the average score of the intensity and distress scale across all intrusions, whilst higher values indicate higher intensity/distress of reported intrusions.

SECONDARY OUTCOMES:
Distress caused by the trauma film: Impact of Event Scale-Revised (IES-R) | At the follow-up measurement (7 days after the experimental manipulation).
  Participants are asked to respond 22 items in reference to the trauma film (e.g., "Pictures about the film popped into my mind.") by indicating how often each reaction occurred during the past seven days with respect to the film they watched last week. Items are rated on a 4-point-Likert-scale ranging from 0 ("not at all"), 1 ("rare"), 3 ("sometimes") to 5 ("often"). The IES-R consists of three subscales: "intrusion", "hyperarousal", and "avoidance". The total score (sum score for the total scale comprising the sum scores of all three subscales) is calculated ranging from 0 to 110 with higher values represent a worse outcome, i.e., higher total distress due to the trauma film in the past week. In addition, the sum score for the intrusion subscale is separately calculated ranging from 0 to 35 (Items 1, 3, 6, 9, 14, 16, 20) with higher values represent more intrusions due to the trauma film in the past week.
Laboratory assessment of intrusive memories: Intrusion Provocation Task (IPT) | At the follow-up measurement (7 days after the experimental manipulation).
  In the Intrusion Provocation Task (IPT), participants are presented with a ten-second long neutral still image from each of the film clips. Immediately afterwards for the next two minutes, they are allowed to think freely and report intrusions by raising a finger. The investigator counts how often the participant lifts his finger in the two minutes. The IPT intrusion score is calculated by the total frequency of intrusions, whilst higher values represent more intrusions.

OTHER OUTCOMES:
Appraisals of Intrusions Questionnaire | At baseline and the follow-up measurement (7 days after the experimental manipulation).
  The Appraisals of Intrusions Questionnaire is 25-item measure that assesses metacognitions of intrusive thoughts and memories. Participants rated the strength of each belief when they experienced their intrusive memories on a scale ranging from 0 (I didn't believe that at all.) to 100 (I was completely convinced that this was true.). Metacognitive appraisals are divided into four categories: "necessity of control", "external consequences", "psychological problem" and "negative self-evaluation". A total score is calculated, whilst higher values indicate more dysfunctional metacognitive beliefs.
Retrospective Assessment of Active Processing | At the follow-up measurement (7 days after the experimental manipulation) retrospectively on Days 1 to 7 after the experimental manipulation.
  Participants are asked in a self-report questionnaire to report for each day and each film clip the amount of time they spent actively processing the content of the film or intrusions associated to it, e.g., by intentionally thinking about it or by discussing it with other people. The participants are asked to rate how many minutes each day they have consciously dealt with the specific film clips or the memories of them. The scale ranges from 0 to 100 minutes in order to pre-define a lower and upper bound. The total score is calculated, whilst higher values indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Lotta Brakemeier, Professor, Principal Investigator — Philipps University Marburg; Winfried Rief, Professor, Principal Investigator — Philipps University Marburg
Locations (1):
- Division of Clinical Psychology and Psychological Interventions, Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Holmes EA, Bourne C. Inducing and modulating intrusive emotional memories: a review of the trauma film paradigm. Acta Psychol (Amst). 2008 Mar;127(3):553-66. doi: 10.1016/j.actpsy.2007.11.002. Epub 2008 Jan 29. PMID 18234153
- [Background] James EL, Lau-Zhu A, Clark IA, Visser RM, Hagenaars MA, Holmes EA. The trauma film paradigm as an experimental psychopathology model of psychological trauma: intrusive memories and beyond. Clin Psychol Rev. 2016 Jul;47:106-42. doi: 10.1016/j.cpr.2016.04.010. Epub 2016 Apr 21. PMID 27289421
- [Background] Iyadurai L, Visser RM, Lau-Zhu A, Porcheret K, Horsch A, Holmes EA, James EL. Intrusive memories of trauma: A target for research bridging cognitive science and its clinical application. Clin Psychol Rev. 2019 Apr;69:67-82. doi: 10.1016/j.cpr.2018.08.005. Epub 2018 Aug 23. PMID 30293686